CLINICAL TRIAL: NCT02174055
Title: Identifying and Measuring Depression in Older Cancer Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Fordham University (Other)
Responsible Party: Sponsor
Other Study IDs: 14-101
Record Dates: First submitted 2014-06-20; First posted 2014-06-25 (Estimated); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Older Cancer Patients
Keywords: Depression; 14-101
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cancer Patients: This protocol aims to design, develop and pilot test a psychometric assessment for depression in older cancer patients. The study is divided in three phases. In Phase 1, approximately 15 depressed patients (as determined clinically) and approximately 15 non-depressed patients will undergo individual interviews. In Phase 2, the team will use the themes and subthemes obtained in Phase 1 to write a set of indicators into questionnaire form. In Phase 3, the newly developed questionnaire will be given to a sample of approximately 150 cancer patients who meet the eligibility criteria. Survey results obtained from this sample of 150 patients will be used to assess internal consistency, conduct item analysis, and determine the unique content of the proposed instrument.
  Interventions: Behavioral: Patient Interviews; Behavioral: newly developed questionnaire; Behavioral: Pilot Testing the Draft Measure

INTERVENTIONS:
Behavioral: Patient Interviews — participate in a brief interview
Behavioral: newly developed questionnaire — 10-16 patients will review draft items and participate in a cognitive interview. 15 older patients will complete the draft measure in order to generate preliminary psychometric data. All interviews will be audio recorded and transcribed by Ubiqus Transcription Company. The audio recordings are uploaded through Ubiqus's secure server and the transcribed audio is returned to the research staff within 48 hours.
Behavioral: Pilot Testing the Draft Measure — The draft measure (approximately 35 items, described above) will be administered to a large sample of older cancer patients (n=150) to generate data to evaluate preliminary psychometric properties (item properties including measures of central tendency, skewness/kurtosis, internal consistency, test/re-test reliability, and construct validity (i.e, convergent and discriminant).and known group differences) to further winnow the measure to include approximately 20 items.

SUMMARY:
The purpose of this study is to develop an accurate and useful way of measuring older patients' moods and reactions to the combined issue of cancer treatment and aging. Also, the purpose of this study is to test a new self-report measure of depressive symptoms tailored to the needs of older adults with cancer. Findings from this research will help us develop improved methods of diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

For Patients in Phases 1- 3:

* Current or previous cancer diagnosis and treatment (any site and any stage)
* All Phases 1,2,3- 70 years of age or older
* For Phase 1b only; 50 participants ages 50-69 will also be recruited
* For Phase 2 only: As per medical record or self report, history of Depression, Dysthymia, or Adjustment Disorder with Depressed Mood
* For Phase 3 depressive subset: As per medical record or self report, a history of depressive symptoms such as

  * Adjustment Disorder with depressed mood
  * Adjustment Disorder with mixed depressed mood and anxiety
  * Mood disorder (i.e., due to general medical condition, Not Otherwise Specified)
  * Depressive Disorder (i.e., Major Depressive Disorder (MDD) single episode, MDD recurrent, Depressive disorder not otherwise specified, Dysthymia)
* In the judgment of the consenting professional able to communicate, comprehend, and complete questionnaires in English

Exclusion Criteria:

For Patients in Parts 1- 3:

* In the judgment of the consenting professional and/or as per medical record, severe psychopathology or cognitive impairment likely to interfere with the participation or completion of the protocol or ability to provide meaningful information.
* For Phase 1&2 only: Score of > 11 on the Blessed Orientation-Memory-Concentration Scale (BOMC)
* For Part 2 only: As per medical record or self report, a diagnosis of a Schizophrenia Spectrum Disorder, current substance use disorder, Bipolar Disorder or Schizotypal personality disorder. Schizophrenia Spectrum Disorders include Schizophrenia, Schizophreniform disorder, Schizoaffective disorder, Delusional disorder, Brief psychotic disorder, Attenuated Psychotic Disorder, and Adjustment Disorder (except for Adjustment Disorder with Depressed Mood).

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: For all Phases, patients who are identified as eligible will be approached in-person in the outpatient clinics or the MSK Counseling Center by members of the research staff, or by letter (physical or electronic).
Sampling Method: Non-Probability Sample
Enrollment: 329 (Estimated)
Dates: Start 2014-06-20 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
develope psychometric assessment of a self report measure of depression | 2 years
  This protocol aims to design, develop and pilot test a psychometric assessment for depression in older cancer patients.
identify differences in item endorsement between younger and older cancer patients on existing depression measures. | 1 year
  These participants will be asked to complete several existing depression measures.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Nelson, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/